CLINICAL TRIAL: NCT03749941
Title: Safety of EUS-FNA for Pancreatic Solid-Pseudopapillary Neoplasm (SPN) Before Surgical Resection: An European Multicenter Registry-based Study on 149 Patients
Brief Title: Safety of EUS-FNA for Pancreatic Solid-Pseudopapillary Neoplasm (SPN) Before Surgical Resection: the SPN-GRAPHE Series
Acronym: SPN-GRAPHE
Status: Completed | Type: Observational
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, KARSENTI, principal investigator, Société Française d'Endoscopie Digestive
Other Study IDs: 2018-SPN-GRAPHE
Record Dates: First submitted 2018-11-18; First posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Solid Pseudopapillary Tumor
Keywords: EUS-FNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Solid-pseudopapillary neoplasm (SPN) is a rare type of pancreatic neoplasm. A cytopathological diagnosis is often mandatory before performing surgical resection. Endo-ultrasonography with fine needle aspiration (EUS-FNA) improve significantly pre-operative SPN diagnosis accuracy. So far, few EUS-FNA performed for SPN were published, and safety of EUS-FNA for SPN has never been investigated. This retrospective European multicenter case-control study compared the recurrence rate in patients with and without EUS-FNA performed before primary tumor resection.

DETAILED DESCRIPTION:
This European multicenter study was conducted in 22 digestive units from the GRAPHE (French taskforce of gastroenterologists working on digestive endoscopy: Groupe de Réflexion et d'Action des Praticiens Hépatogastroentérologues en Endoscopie Digestive), and retrospectively included all patients who have undergone complete resection of their pancreatic SPN from 2000 to 2018. The use of the diagnostic filing software of each unit of cytopathology, endoscopy and digestive surgery allowed the completeness of the prospection in each center.

The data were retrospectively collected by extraction from our medical patient management softwares.

The following data were collected: age, gender, symptoms, tumor size, tumor location (uncus, head, isthmus, body or tail of the pancreas), presence of tumor calcifications, performing of a EUS-FNA for diagnostic purposes before surgical resection, follow-up, and diagnosis of recurrence of the SPN during follow-up. Other data were collected in case of EUS-FNA: path of the needle puncture (transgastric or transduodenal), diameter of the needle, number of passes, immediate EUS-FNA morbidity, and EUS-FNA diagnosis of SPN (certain, probable, false or absent).

Patients with and without initial EUS-FNA were compared and the main criteria of this study was determinate: the presence of recurrence of the SPN during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients who have undergone complete resection of their pancreatic SPN were included. Inclusion criterion was the definite diagnosis of SPN on the pathological examination of the complete tumor resection specimen.

Exclusion Criteria:

* No

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This European multicenter study was conducted in 22 digestive units from the GRAPHE (French taskforce of gastroenterologists working on digestive endoscopy: Groupe de Réflexion et d'Action des Praticiens Hépatogastroentérologues en Endoscopie Digestive), and retrospectively included all patients who have undergone complete resection of their pancreatic SPN from 2000 to 2018. The use of the diagnostic filing software of each unit of cytopathology, endoscopy and digestive surgery allowed the completeness of the prospection in each center.
  The data were retrospectively collected by extraction from our medical patient management softwares.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Recurrence after primary tumor resection | through study completion, an average of 43 months
  Recurrence after primary tumor resection confirmed during follow up